CLINICAL TRIAL: NCT06850571
Title: Evaluation of the Clinical Outcomes and Cost-effectiveness of Aflibercept and Bevacizumab in Iraqi Patients With Diabetic Maculopathies: Open Label Parallel Groups Clinical Trial
Brief Title: Aflibercept and Bevacizumab for Diabetic Maculopathies
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Collaborators: Baghdad Medical City (Other)
Responsible Party: Principal Investigator, Mohammed Mahmood Mohammed, Principal Investigator, Al-Mustansiriyah University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOM4540
Record Dates: First submitted 2025-02-15; First posted 2025-02-27 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Maculopathy
MeSH Terms: interventions — Bevacizumab; Injections; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab group (Active Comparator): Patients will receive an intravitreal injection of 1.25 mg (in 0.05 ml solution) of bevacizumab once monthly for three consecutive months.
  Interventions: Drug: Bevacizumab Injection [Avastin]
- Aflibercept group (Experimental): Patients will receive an intravitreal injection of 2.0 mg (in 0.05 ml solution) of aflibercept once monthly for three consecutive months.
  Interventions: Drug: Aflibercept 2Mg/0.05Ml Inj,Oph

INTERVENTIONS:
Drug: Bevacizumab Injection [Avastin] — 1.25 mg intravitreal injection given once monthly for three consecutive months.
  Other Names: Avastin 100 mg in 4 ml Injection
  Arms: Bevacizumab group
Drug: Aflibercept 2Mg/0.05Ml Inj,Oph — 2.0 mg intravitreal injection given once monthly for three consecutive months.
  Other Names: EYLEA Bayer
  Arms: Aflibercept group

SUMMARY:
The goal of this clinical trial is to to evaluate the clinical outcomes following treatment with bevacizumab versus aflibercept. These outcomes include:

* Functional changes: The visual outcomes achieved by testing visual acuity
* Anatomical changes: macular thickness and edema by optical coherence tomography (OCT).

DETAILED DESCRIPTION:
Brief summary template The goal of this clinical trial is to to evaluate the clinical outcomes following treatment with bevacizumab versus aflibercept. These outcomes include:

* Functional changes: The visual outcomes achieved by testing visual acuity
* Anatomical changes: macular thickness and edema by optical coherence tomography (OCT).

The secondary objectives include:

* Analyze the cost-effectiveness of bevacizumab versus aflibercept in the management of diabetic maculopathies.
* Safety profile and adverse events reported with bevacizumab and aflibercept use and their association with changes functioning changes

Patients inclusion criteria include patients both sexes, age over 40 years with type 2 diabetes mellites diagnosed with diabetic maculopathies; those patients with reduced or reducing vision (6/9-6/90) according to visual acuity and significant foveolar thickening on OCT (more than 250 μm).

Researchers will compare patients with intravitreal anti-VEGF treatment, aflibercept or bevacizumab for three successive monthly injections to see if there are any differences in safety and efficacy between the two arms.

Participants will take aflibercept or bevacizumab intravitreally every month for 3 months

Visit the clinic once every 1 month for checkups and assessment the pre- and post- 3 month anti-VEGF treatment values and findings by:

* Pneumotonometry will be used to measure intraocular pressure (IOP)
* Central foveal thickness (CFT) will be measured by optical coherence tomography (OCT).
* Visual acuity (by Snellen visual acuity chart) will be assessed.
* Pretreatment serum VEGF levels and 7-days after the third anti-VEGF dose

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellites.
* Patients diagnosed with diabetic maculopathies, including focal and diffuse maculopathies, according to Early Treatment of Diabetic Retinopathy Study (ETDRS) criteria
* Patients with reduced or reduced vision (6/9-6/90) according to visual acuity and significant foveolar thickening on OCT (more than 250 μm)
* Patients will be treated with intravitreal anti-VEGF treatment, aflibercept, or bevacizumab for three successive monthly injections.

Exclusion Criteria:

* Patients with type 1 diabetes mellites
* Patients with type 2 on insulin therapy.
* Patients who were previously treated with intravitreal anti-VEGF within the previous three months or intravitreal corticosteroids for six months
* Prior macular photocoagulation or photodynamic therapy, prior intraocular surgeries within three months (laser & surgery may cause edema)
* Pregnant or nursing women
* In patients with a history of thromboembolic events, systemic VEGF inhibition is likely to cause cardiovascular complications, such as arterial thromboembolic events.
* Patients major surgery within the previous one year or planned within the next few months that may interfere with anti-VEGF treatment
* Uncontrolled hypertension as hypertension is associated with the use of VEGF antagonists.
* Known coagulation abnormalities or current use of anticoagulative medication other than aspirin.
* Hemorrhagic macular infarction is reported with the use of VEGF antagonists.
* Patients with intraocular pressure more than 25 mmHg
* Presence of iris neovascularization/vitreous hemorrhage

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual accuty assessed by snellen chart | one day before start of treatment, and after 3 months of starting the treatment
  The visual outcomes achieved by testing visual acuity by snellen chart
Central fovial thinkness by OCT | one day before start of treatment, and after 3 months of starting the treatment
  Macular thickness by optical coherence tomography (OCT)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | During the three months after starting the treatment till the end of follow-up.
  Safety profile and adverse events reported Safety profile and adverse events reported with bevacizumab and aflibercept use and their association with changes in functioning changes.
Quality of life assessed by Visual Functioning Questionnaire 25 (ARB-VFQ-25) | one day before start of treatment, and after 3 months of starting the treatment
  Quality of life-related to visual functioning will be assessed using the Arabic version of the Visual Functioning Questionnaire 25 (ARB-VFQ-25). The ARB-VFQ-25 will be assessed and validated before the start of data collection.
Adherence assessed by Adherence Barriers Questionnaire of Intravitreal Therapy (ABQ-IVT) | one day before start of treatment, and after 3 months of starting the treatment
  Assessment and validation of the Arabic version of the Adherence Barriers Questionnaire of Intravitreal Therapy (ABQ-IVT) and studying the barriers to adherence that may affect intravitreal drug use.

CONTACTS AND LOCATIONS:
Locations (1):
- Baghdad Medical City Complex, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided